CLINICAL TRIAL: NCT01699958
Title: A Pilot Study of the "Healthy Living Study," a Randomized Controlled Trial of a Brief Outpatient Problem-solving Intervention to Promote Healthy Eating and Activity Habits in Adolescents.
Brief Title: A Brief Outpatient Problem-solving Intervention to Promote Healthy Eating and Activity Habits in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: StanfordIRB-20922; T32MH019938 (NIH)
Record Dates: First submitted 2012-09-28; First posted 2012-10-04 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-10

CONDITIONS: Health Behavior
Keywords: Problem solving therapy; Behavior change
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Problem-solving intervention (Experimental): 2 individual sessions teaching problem-solving skills with the use of videos, handouts, and worksheets.
  Interventions: Behavioral: Problem-solving intervention
- Control: Standard Care (No Intervention): Control arm participants will receive standard of care from their primary care provider.

INTERVENTIONS:
Behavioral: Problem-solving intervention — Participants will receive 2 individual sessions teaching and reviewing problem-solving skills.
  Arms: Problem-solving intervention

SUMMARY:
The purpose of this study is to refine, evaluate the feasibility, and to estimate the effect of the "healthy Living Study," a brief outpatient problem-solving intervention to promote healthy eating and activity habits in adolescents.

DETAILED DESCRIPTION:
This study will refine, evaluate the feasibility, and estimate the effect of a brief problem-solving intervention to promote healthy eating and activity habits in adolescents. Intervention participants will receive 2 sessions of individual behavioral counseling on problem-solving skills utilizing educational videos, handouts, and worksheets. Intervention participants will be asked to generate unique health goals and practice utilizing problem-solving skills to achieve these goals.Control participants will receive standard of care. Outcomes will explore the ability to shorten the intervention, integrate the intervention into busy outpatient clinics, and estimate the effect of the intervention on confidence to maintain or improve healthy habits and to improve problem-solving skills.

ELIGIBILITY:
Inclusion Criteria:

* 13-18 years old
* Able to read and speak English
* Patient of the Lucile Packard Children's Hospital teen clinic, weight clinic, or mobile teen van

Exclusion Criteria:

* History of purging within the prior 12 months

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2011-06; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Feasibility to conduct a brief problem-solving intervention in a busy academic outpatient setting. | From recruitment of the first participant to completion of the intervention by the last participant, anticipated duration of time: 7-8 months
  Feasibility will be measured in the following ways:
  1. Refinement of the intervention by the end of the study to a reasonable length to compliment average patient clinic visits with a goal of 30 minutes or less
  2. Minimal disruption of clinic flow measured through clinic provider and staff satisfaction surveys and qualitative comments during the course of the intervention

SECONDARY OUTCOMES:
Change in problem-solving skills | Change from baseline to 1-2 months
  Participants will complete survey questions modified from the Social Problem-Solving Inventory for Adolescents (SPSI-A) both pre-intervention and post-intervention. These questions provide an assessment of problem-solving skills and are scored on a Likert scale of 1-5 with 5=more positive/constructive problem-solving skills. Change in overall mean score from pre- to post- intervention will be compared within intervention and control groups and between groups. Duration of time between pre- and post- intervention will average 1-2 months.
Change in confidence to maintain or improve healthy eating habits | Change from baseline to 1-2 months
  Participants will complete pre- and post- intervention questions on confidence to maintain or improve healthy eating habits. An example question: "How confident are you that you could change or maintain your eating patterns to limit soda to <1 can/day." Questions will be scored on a Likert scale of 1-6 with 6=very confident. Change in overall mean score from pre- to post- intervention will be compared within intervention and control groups and between groups. Duration of time between pre- and post- intervention will average about 1-2 months.
Sufficient recruitment and retention rates | From recruitment of the first participant to completion of the intervention by the last participant, anticipated duration of time: 7-8 months
  Detailed records of patients approached, consented, randomized, and completing the study will be maintained. These records will be reviewed at the conclusion of the study to gauge patient interest in participating in a problem-solving intervention in the outpatient setting.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Gee, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Palo Alto, California, United States